CLINICAL TRIAL: NCT01699074
Title: Acute Dose Response Effects of Korean White Ginseng (Panax Ginseng C.A. Meyer) on Cardiovascular Disease Risk Factors in Individuals With Metabolic Syndrome or Type 2 Diabetes
Brief Title: Acute Dose Response of Korean White Ginseng in Metabolic Syndrome or Type 2 Diabetes
Acronym: KWG
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 182629
Record Dates: First submitted 2012-10-01; First posted 2012-10-03 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-04

CONDITIONS: Type 2 Diabetes; Metabolic Syndrome
Keywords: Korean White Ginseng; Type 2 diabetes; Metabolic syndrome
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Metabolic Syndrome | interventions — Asian ginseng

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- 1 gram of White Korean Ginseng (Experimental): 1 gram of White Korean Ginseng
  Interventions: Dietary Supplement: 1 gram of White Korean Ginseng
- 3 grams of White Korean Ginseng (Experimental): 3 grams of White Korean Ginseng
  Interventions: Dietary Supplement: 3 grams of White Korean Ginseng
- 6 grams of White Korean Ginseng (Experimental): 6 grams of White Korean Ginseng
  Interventions: Dietary Supplement: 6 grams of White Korean Ginseng
- 3 grams of Wheat Bran Control (Placebo Comparator): 3 grams of Wheat Bran Control
  Interventions: Dietary Supplement: 3 grams of Wheat Bran Control
- 500mg of Korean Red Ginseng (Active Comparator): 500mg of Korean Red Ginseng
  Interventions: Dietary Supplement: 500mg of Korean Red Ginseng

INTERVENTIONS:
Dietary Supplement: 1 gram of White Korean Ginseng — 1 gram of White Korean Ginseng
  Arms: 1 gram of White Korean Ginseng
Dietary Supplement: 3 grams of White Korean Ginseng — 3 grams of White Korean Ginseng
  Arms: 3 grams of White Korean Ginseng
Dietary Supplement: 6 grams of White Korean Ginseng — 6 grams of White Korean Ginseng
  Arms: 6 grams of White Korean Ginseng
Dietary Supplement: 3 grams of Wheat Bran Control — 3 grams of Wheat Bran Control
  Arms: 3 grams of Wheat Bran Control
Dietary Supplement: 500mg of Korean Red Ginseng — 500mg of Korean Red Ginseng
  Arms: 500mg of Korean Red Ginseng

SUMMARY:
The study is a Phase-I like double blind randomized placebo controlled crossover design trial. The objective is to assess the dose response relationship on glycemic and vascular effects of an acutely administered Korean White Ginseng (KWG)(Panax C.A. Meyer) in individuals with metabolic syndrome or type 2 diabetes . Twenty seven subjects with Type 2 Diabetes (Key inclusion criteria: HbA1c ≤8.5%)or metabolic syndrome (Key inclusion criteria: as defined by The US National Cholesterol Education Program Adult Treatment Panel III)will be recruited for the study.

DETAILED DESCRIPTION:
This study hypothesizes that KWG will dose dependently lower postprandial area under the curve compared to negative control, as well as will dose dependently decrease postprandial glycemia. It also assumes that use of KWG will dose dependently decrease aortic and brachial blood pressure, aortic augmentation index, and mean arterial pressure, and improve left ventricular ejection duration(ED) and subendocardial viability ratio (SEVR) compared to control. Finally, it expects to notice an effect on subjective satiety levels and have no significant adverse effects compared to control.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* 18-75 years old
* BMI 25-35 kg/m2
* Presence of type 2 diabetes (as defined by HbA1c ≤8.5%),treatment with diet or oral hypoglycemic medication) OR
* Presence of Metabolic Syndrome as defined by The US National Cholesterol -Education Program Adult Treatment Panel III (NCEP III). As per NCEP III criteria, at least three of the following must be present:
* central obesity: waist circumference ≥ 102 cm or 40 inches (male), ≥ 88 cm or 36 inches(female)
* dyslipidemia: TG ≥ 1.7 mmol/L (150 mg/dl);
* dyslipidemia: HDL-C < 40 mg/dL (male), < 50 mg/dL (female) blood pressure ≥ 130/85 mmHg; fasting plasma glucose ≥ 6.1 mmol/L (110 mg/dl)

Exclusion Criteria:

* BMI >35 kg/m2
* Hypertensive (brachial systolic BP ≥140mmHg and/or diastolic BP ≥90mmHg)
* Pregnant women, or those at risk of pregnancy, or breastfeeding at the time of the study.
* Women of childbearing age that do not use acceptable method of birth control (ie. abstinence, implants, injectables, oral contraceptives, IUDs etc).
* Chronic conditions including: liver disease, cancer, heavy alcohol use, bleeding disorders, history of angina, congestive heart failure, coronary revascularization, peripheral vascular disease, retinopathy, kidney disease or coronary/cerebrovascular event; chronic use of medications including blood-thinners, SSRIs, MAO inhibitors, medications affecting NO synthesis (eg. Viagra)
* Allergy or sensitivity to the placebo (wheat bran), ginseng or gelatin used in the capsules.
* Use of any ginseng products within three days preceding the study and during the study.
* Allergies to Panax species, their constituents or to other members of the Araliaceae family.

The use of additional NHPs that may affect blood pressure or blood glucose Individuals suffering from glucose-galactose malabsorption syndrome.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-05; Primary Completion 2013-09 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Effect of KWG on vascular and glycemic measures | 3 hours
  To evaluate the acute dose response effect of KWG on blood glucose Area under the Curve (AUC) compared to controls in individuals with Metabolic syndrome or Type 2 Diabetes To evaluate the acute effect of KWG treatments on arterial stiffness as measured by aortic augmentation index (AIx)

SECONDARY OUTCOMES:
Effect of KWG on vascular and glycemic measures | 4 hours
  To evaluate the acute effect of Korean White ginseng treatments on peak and postprandial glycemia measures.To evaluate the acute effect of KWG treatments on aortic and brachial blood pressure To evaluate the acute effect of KWG treatments on heart rate, mean arterial pressure, left ventricular ejection duration (ED) and subendocardial viability ratio (SEVR) - a surrogate marker of myocardial perfusion

OTHER OUTCOMES:
KWG and satiety | 4 hours
  To evaluate the acute effect of KWG treatments on subjective satiety scores to determine any potential effects on appetite control mechanisms compared to controls. Symptoms questionnaire will assess potential adverse effects of treatments (safety)

CONTACTS AND LOCATIONS:
Locations (1):
- : Clinical Nutrition and Risk Factor Modification Centre, St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Shishtar E, Jovanovski E, Jenkins A, Vuksan V. Effects of Korean White Ginseng (Panax Ginseng C.A. Meyer) on Vascular and Glycemic Health in Type 2 Diabetes: Results of a Randomized, Double Blind, Placebo-controlled, Multiple-crossover, Acute Dose Escalation Trial. Clin Nutr Res. 2014 Jul;3(2):89-97. doi: 10.7762/cnr.2014.3.2.89. Epub 2014 Jul 29. PMID 25136536